CLINICAL TRIAL: NCT02431507
Title: Magnetic Apnea Prevention (MAGNAP) Device to Treat Obstructive Sleep Apnea: First-In-Human Study of Feasibility and Safety
Brief Title: Magnetic Apnea Prevention(MAGNAP) Device to Treat Obstructive Sleep Apnea:First-In-Human Study of Feasibility and Safety
Acronym: MAGNAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Michael Harrison (Other)
Responsible Party: Sponsor-Investigator, Michael Harrison, Principal Investigator/ Sponsor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-15689
Record Dates: First submitted 2015-04-23; First posted 2015-05-01 (Estimated); Last update posted 2026-01-22 (Actual); Status verified 2025-12

CONDITIONS: Obstructive Sleep Apnea
Keywords: apnea; sleep apnea; magnetic sleep apnea device; hyoid bone
MeSH Terms: conditions — Sleep Apnea, Obstructive; Apnea; Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment Arm with Magnetic Apnea Device (Experimental): The treatment arm with magnetic apnea device includes: surgical implantation of the magnetic apnea device(MAGNAP) to treat obstructive sleep apnea in each eligible enrolled subject . A custom fitted external brace will be created for wear throughout the 13 months of treatment and evaluated for improvement of symptoms..
  Interventions: Device: Magnap

INTERVENTIONS:
Device: Magnap — This is a non-randomized clinical trial.Patients 21-70 years diagnosed with moderate to severe obstructive sleep apnea will have the Magnap Magnetic Apnea Device surgically implanted on the subject's hyoid bone and used in conjunction with an external neck brace and magnet to open airway during sleep in treatment of Obstructive Sleep Apnea. We will monitor for safety, brace compliance and improvement of symptoms of sleep apnea for a total of 13 months.
  Other Names: Magnetic apnea device

SUMMARY:
The purpose of this study is to determine the safety and feasibility of the Magnap magnetic device in the treatment of obstructive sleep apnea (OSA).

DETAILED DESCRIPTION:
Magnap is a magnet-activated treatment for obstructive sleep apnea (OSA) designed to be less invasive than reconstructive surgery, more tolerable than positive airway pressure, and more effective than non-invasive therapies for OSA. The Magnap device consists of a neodymium-iron-boron rare earth magnet with a ferromagnetic directional back-plate encased in titanium. The device will be implanted surgically on the hyoid bone. Following surgery, the patient is fitted with a custom, removable external neck accessory containing a second magnet, which is worn during sleep and prevents airway collapse by attracting the internal hyoid magnet with sufficient force to keep the airway open .

ELIGIBILITY:
Inclusion Criteria:

* Patient is between 21 and ≤70 years of age
* Subject has moderate to severe obstructive sleep apnea (defined as apnea-hypopnea index of 15-50 events/hour on baseline/screening polysomnogram)
* Subject is intolerant of positive airway pressure therapy (defined as <2 hours of sleep time with use per night for at least 5 nights per week as measured objectively by evaluation of continuous positive airway pressure (CPAP) machine memory chip and interpreted by the study sleep medicine specialist)
* Subject signs and dates a written informed consent form and indicates understanding of the study procedures and risks

Exclusion Criteria:

* Any evidence that apnea is not caused by base of tongue (i.e., central apnea, neurologic disorder, retropalatal collapse, nasal obstruction)
* Any condition likely requiring MRI or has a metal implant
* Any factor that, in the surgeon's judgment, would pose a risk to surgery or placement of a long-term implanted device
* Any factor that, in the surgeon's judgment, would make the subject unlikely to respond to Magnap treatment
* Congenital anomalies of the larynx, pharynx, or trachea or any other anatomical abnormality of the head, neck, or chest that would be a contraindication to placement of the Magnap device and usage of the external device
* There are no exclusion criteria based on gender, race or ethnicity

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-09; Primary Completion 2026-12-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Ability of the subject to use the Magnap device for the duration of the study. | 13 months
  Determined by: monitoring for successful device implantation without complications necessitating device removal in all 10 subjects, subjects able to use the device throughout study period once fitted with the brace. Safety will be monitored by tracking all adverse events in 10 subjects and/or complications of treatment.

SECONDARY OUTCOMES:
Ability of external device to open the airway, | 13 Months
  Outcomes will be measured by pharyngeal airway measurements taken pre and post implantation with and without the external device and recording improvements of OSA parameters recorded on polysomnogram pre and post-implantation with and without the external device.
Improve symptoms related to OSA | 13 Months
  Measurement of symptom improvement and compliance will be monitored by questionnaires 4 times during the study and by 4 polysomnograms after implantation. All 10 subjects will be required to complete daily or event journal entries describing changes and/or experiences with the brace and OSA symptoms
Measure Patient compliance | 13 Months
  Measurement of symptom improvement will be documented and compared to all post-implantation polysomnograms and compliance will be monitored by daily sleep journal entries by all subjects.questionnaires and journal entries.

CONTACTS AND LOCATIONS:
Overall Officials: Michael R Harrison, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco/Mount Zion Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosenbluth KH, Kwiat DA, Harrison MR, Kezirian EJ. Hyoid bone advancement for improving airway patency: cadaver study of a magnet-based system. Otolaryngol Head Neck Surg. 2012 Mar;146(3):491-6. doi: 10.1177/0194599811429522. Epub 2011 Nov 22. PMID 22114308